CLINICAL TRIAL: NCT00727844
Title: A Phase 2a, Randomized, 2-Arm, Open-Label, Clinical Trial of the Efficacy of Linezolid Combined With Antituberculous Therapy in Subjects With Extensively Drug-Resistant (XDR) Pulmonary Tuberculosis
Brief Title: Linezolid to Treat Extensively-Drug Resistant Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Clifton E. Barry III, Ph.D., Principal Investigator, Tuberculosis Research Section (TRS), National Institute of Allergy and Infectious Diseases (NIAID)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-I-N167
Record Dates: First submitted 2008-08-01; First posted 2008-08-04 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Tuberculosis; Multidrug Resistant Tuberculosis; Extensively Drug Resistant Tuberculosis
Keywords: XDR-TB; Linezolid; Drug Resistance; Computed Tomography; Pharmacokinetics; Tuberculosis; Drug Resistance Tuberculosis; MDR-TB
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis; Tuberculosis | interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delayed Start Linezolid (Experimental): Subjects continued their existing regimen for 2 months after which LZD (600 mg once daily) was added. After 2 consecutive AFB negative sputum smears (not to exceed 4 months of LZD therapy), subjects were randomized to continue on 600 mg LZD once daily or to de-escalate to 300 mg once daily. Regardless of the dosage, subjects remained on LZD treatment for 18 months after sputum culture conversion or until they could no longer tolerate therapy.
  Interventions: Drug: Delayed Start Linezolid
- Immediate Start Linezolid (Experimental): Upon completion of entry criteria, subjects had LZD (600 mg once daily) added to their regimen. After 2 consecutive AFB negative sputum smears (or at 4 months) subjects were randomized to continue on 600 mg LZD once daily or to de-escalate to 300 mg once daily. Regardless of the dosage, subjects remained on LZD treatment for 18 months after sputum culture conversion or until they could no longer tolerate therapy.
  Interventions: Drug: Immediate Start Linezolid

INTERVENTIONS:
Drug: Immediate Start Linezolid
  Other Names: Zyvox
  Arms: Immediate Start Linezolid
Drug: Delayed Start Linezolid
  Other Names: Zyvox
  Arms: Delayed Start Linezolid

SUMMARY:
This study, conducted in Masan and Seoul, South Korea, investigated the effectiveness of linezolid (LZD) in treating patients with extensively drug resistant tuberculosis (XDR TB). Because regular medicines do not work well against XDR TB, many more people die from it than from regular TB, which can be successfully treated by taking TB medication for 6 months. Linezolid has been used to treat other kinds of infections, but has not been well studied for TB. This study examined the side effects and effectiveness of prolonged treatment with linezolid at two different doses.

People 20 years of age and older who have XDR TB were eligible for this 3-year study.

Participants underwent the following tests and procedures:

* LZD treatment: Patients were randomly assigned to one of two study groups. Group 1 patients were observed for 2 months before starting LZD, while group 2 patients begin taking LZD right away. Both groups began with a 600 mg daily dose of LZD. After patients stopped coughing up TB germs (or after 4 months on LZD) they were randomly assigned either to continue taking 600 mg of LZD for the rest of the study or to take a decreased dose of 300 mg. In addition to LZD, patients continued to take their currently prescribed TB medications.
* Medical history.
* Physical examinations each month during treatment.
* Sputum collections once a week or more until 3 weeks after the patient was no longer contagious.
* Blood draws every week for 16 to 24 weeks and then once a month.
* Urine collections at several time points.
* Nerve and eye examinations before starting treatment and then monthly to look for possible LZD side effects.
* CT scans of the lungs three to four times the first year and once more later in the study. For this test the patient lay on a table within the doughnut-shaped CT scanner while special X-ray pictures are taken.

Patients who participated in a substudy had PET scans instead of the CT scans. For this test, the patient was given an injection into a vein of a radioactive chemical that can be detected by a special camera and viewed on a screen. The patient lay on a table within the doughnut-shaped scanner while pictures were taken.

DETAILED DESCRIPTION:
World-wide, there is an increasing incidence of multi-drug resistant tuberculosis (MDR-TB) and extensively drug-resistant TB (XDR-TB). For patients diagnosed with either of these deadly diseases, effective drug treatment options are sub-optimal or non-existent. In South Korea, there are a growing number of patients not responding to any therapy who have little hope for survival without new drugs. Linezolid (LZD), an antimicrobial approved for gram positive bacterial infections, has been used off-label for drug resistant TB and is quickly becoming a sought after drug for this population, despite lack of clinical evidence of efficacy. At the present time the prohibitive cost of LZD limits widespread use; however, when patent exclusivity expires in May of 2015 it will be imperative to have examined the benefits versus risks of LZD for TB in a controlled setting. The National Masan Tuberculosis Hospital (NMTH) in Masan, South Korea and the National Medical Center in Seoul, South Korea provide us with an opportunity to systematically address questions about LZD in a highly drug-resistant population.

This is a Phase 2a, randomized, 2-arm study of LZD, which evaluated the efficacy, safety, and tolerability of LZD in subjects whose isolates have shown resistance to all known active TB drugs or who have failed to respond to any active drugs to which they are susceptible. Subjects were required to have been on a failing regimen for at least 6 months prior to study entry, with persistent sputum smear positivity, culture positivity and no significant clinical sign of response to therapy. To be considered for the study, a subject's treatment plan must have been stable without the addition of drugs to which the subjects isolate was suspected to be sensitive: however drugs may have been discontinued during this time. Subjects were stratified based upon a diagnosis of diabetes mellitus (type I and II included) using block randomization. At the primary randomization, subjects were randomly assigned either to immediately add 600 mg LZD once daily to their existing regimen or to a delay of 2 months before adding 600 mg LZD once daily to their existing regimen. A second randomization occurred after 2 consecutive negative sputum smears or at 4 months after the start of LZD therapy (whichever came first), when subjects either stayed with their current 600 mg LZD once daily or de-escalated to 300 mg LZD once daily (see Section 4.1.4 Study Schema). The second randomization was stratified on diabetes. The primary objective of this study was to evaluate the efficacy of LZD therapy, as measured by sputum culture conversion. Secondary aims of this study included: investigation of the pharmacokinetic and pharmacodynamic profiles of LZD in blood; tolerability and toxicity of prolonged LZD administration at doses of 300 mg and 600 mg daily; the rate of change of radiological findings by computed tomography (CT); the rate of relapse 12 months after discontinuation of therapy; the rate of development of drug resistance to LZD; changes in immunologic and bacterial lipid markers during LZD therapy; the correlation of whole-blood killing assays with response to LZD therapy; and effects of LZD on mitochondrial function, a potential early indicator of LZD toxicity. In a substudy, we aimed to investigate the changes in lung architecture and cellular activity during treatment using F-fluoro-2-deoxy-D-glucose - positron emission tomography-computed tomography (FDG-PET-CT) of 20 subjects on LZD therapy. Estimated total study duration for each subject was approximately 3 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males and females age 20 and above

Documented pulmonary tuberculosis at screening

Radiographic evidence of tuberculous disease of the lung(s)

History of chronic, AFB positive sputum smears and culture positive TB

Mycobacterium species identification as Mycobacterium tuberculosis

Confirmed resistance to INH, RIF, kanamycin, ofloxacin, and moxifloxacin by genotypic or phenotypic testing OR subjects with documented failure to respond to treatment despite DST susceptibility

Failure to respond (after at least 6 months) to a anti-TB drug regimen including any known active agents

Willingness to be an inpatient until 2 consecutive AFB-negative sputum smears

When an outpatient, willing to come back for weekly tests and scheduled follow-up visits

Willingness to have samples stored

Ability and willingness to give written or oral informed consent

EXCLUSION CRITERIA:

Subjects below 20 years of age

Subjects who have previously been on LZD

Women of childbearing potential, who are pregnant, breast feeding, or unwilling to avoid pregnancy (i.e., the use of appropriate contraception including oral and subcutaneous implantable hormonal contraceptives, condoms, diaphragm, intrauterine device (IUD), or abstinence from sexual intercourse). [Note: Prospective female participants of childbearing potential must have negative pregnancy test (urine) within 48 hours prior to study entry.]

Men who are unwilling to use contraceptives or practice abstinence

People with any of the following in their current medical assessments:

Absolute neutrophil count less than 1000 cells/mL

White blood cell count (WBC) less than 3.0 X 10(3)/microL

Hemoglobin less than 7.0 g/dL

Platelet count less than 75,000 cells/mm(3)

Serum creatinine greater than 2.0 mg/dL

Aspartate aminotransferase (AST or SGOT) greater than 100 IU/L

Alanine aminotransferase (ALT or SGPT) greater than 100 IU/L

Total bilirubin greater than 2.0 mg/dL

Moderate or severe peripheral or optical neuropathy (or a history of)

HIV-1 or HIV-2 infection

Systemic lupus erythematosus, rheumatoid arthritis, or other connective tissue disease

Patients who, in the investigator's judgment, are too ill to participate in the study

History of allergy or serious adverse reaction to the LZD formulation used in this study

Patients with anticipated surgical intervention

The use of any of the following drugs within 30 days prior to study or anticipated use of these drugs within the next 60 days: (Please not, bronchodilators and cough syrup (or similar cough medicines) are allowed before and during the study if blood pressure is monitored regularly, per Contraindications, p.12, of the Zyvox Package Insert.)

Selective serotonin reuptake inhibitors (SSRIs)

Monoamine oxidase inhibitors (MAOIs)

Systemic cancer chemotherapy

Systemic corticosteroids

Systemic investigational agents

Antiretroviral medications

Growth factors

HIV vaccines

Immune globulin

Interleukins

Interferons

The need for ongoing therapy with antidepressants (SSRI, MAOI), hydroxyzine, dopaminergic agents (such as Sinemet, dopamine, and dobutamine), lithium, cyclosporine, tacrolimus, sirolimus, and levodopa (such as sinemet) while on study drug

Any other serious systemic illness requiring treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy for at least 14 days prior to study entry

Patients who the physician has reason to believe may have been non-compliant in the previous 12 months of treatment

SUBSTUDY ELIGIBILITY CRITERIA

INCLUSION CRITERIA:

Subjects who meet the inclusion criteria for main study are eligible for the substudy.

EXCLUSION CRITERIA:

Exclusion criteria for main study apply to the substudy with the exception that subjects with uncontrolled diabetes mellitus will be excluded from the substudy. The study physician may decide that a patient is healthy enough to participate in the main study but not the sub-study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-07; Primary Completion 2012-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifton Barry, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- South Korea (2):
  - National Masan Tuberculosis Hospital, Changwon
  - National Medical Center, Seoul

REFERENCES:
- [Background] Richter E, Rusch-Gerdes S, Hillemann D. First linezolid-resistant clinical isolates of Mycobacterium tuberculosis. Antimicrob Agents Chemother. 2007 Apr;51(4):1534-6. doi: 10.1128/AAC.01113-06. Epub 2007 Jan 22. PMID 17242139
- [Background] Hillemann D, Rusch-Gerdes S, Richter E. In vitro-selected linezolid-resistant Mycobacterium tuberculosis mutants. Antimicrob Agents Chemother. 2008 Feb;52(2):800-1. doi: 10.1128/AAC.01189-07. Epub 2007 Dec 10. No abstract available. PMID 18070973
- [Background] Duncan K, Barry CE 3rd. Prospects for new antitubercular drugs. Curr Opin Microbiol. 2004 Oct;7(5):460-5. doi: 10.1016/j.mib.2004.08.011. PMID 15451500
- [Result] Lee M, Lee J, Carroll MW, Choi H, Min S, Song T, Via LE, Goldfeder LC, Kang E, Jin B, Park H, Kwak H, Kim H, Jeon HS, Jeong I, Joh JS, Chen RY, Olivier KN, Shaw PA, Follmann D, Song SD, Lee JK, Lee D, Kim CT, Dartois V, Park SK, Cho SN, Barry CE 3rd. Linezolid for treatment of chronic extensively drug-resistant tuberculosis. N Engl J Med. 2012 Oct 18;367(16):1508-18. doi: 10.1056/NEJMoa1201964. PMID 23075177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study patients recruited from 12/2008 to 5/2011 at the National Masan Hospital, Changwon, Korea and the National Medical Center, Seoul, Korea.
Groups:
- Initial Randomization: Immediate Start Linezolid: Upon completion of entry criteria, subjects immediately added linezolid 600 mg once daily to their ongoing TB treatment regimen.
- Initial Randomization: Delayed Start Linezolid: Subjects continued their existing treatment regimen for 2 additional months after which linezolid 600 mg once daily was added.
- 2nd Randomization: Linezolid 600 mg Daily; 2nd Randomization: Linezolid 300 mg Daily: After conversion to negative sputum smears (or receipt of 4 months of therapy), patients underwent a second randomization, stratified according to diabetes mellitus status, either to continue receiving linezolid at a dose of 600 mg per day or to receive a lower dose, 300 mg per day, for an additional 18 months or until therapy was stopped owing to side effects or laboratory abnormalities.
Period: Initial Randomization
Arm/Group | Initial Randomization: Immediate Start Linezolid | Initial Randomization: Delayed Start Linezolid | 2nd Randomization: Linezolid 600 mg Daily | 2nd Randomization: Linezolid 300 mg Daily
Started | 21 (2 patients withdrawn before receiving any linezolid owing to baseline neuropathy) | 20 | 0 | 0
Included in MITT Analysis | 19 | 20 | 0 | 0
Completed | 19 | 20 | 0 | 0
Not Completed | 2 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Period: Second Randomization
Arm/Group | Initial Randomization: Immediate Start Linezolid | Initial Randomization: Delayed Start Linezolid | 2nd Randomization: Linezolid 600 mg Daily | 2nd Randomization: Linezolid 300 mg Daily
Started | 0 | 0 | 17 (6 patients excluded before 2nd randomization: 2 had withdrawn and 4 already dose reduced due to AE) | 16 (6 patients excluded before 2nd randomization: 2 had withdrawn and 4 already dose reduced due to AE)
Completed | 0 | 0 | 17 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2 patients excluded in immediate start group before receiving any linezolid owing to baseline neuropathy
Groups:
- Immediate Start Linezolid: Upon completion of entry criteria, subjects will have LZD (600 mg once daily) added to their regimen. After 2 consecutive AFB negative sputum smears (or at 4 months) subjects will be randomized to continue on 600 mg LZD once daily or to de-escalate to 300 mg once daily. Regardless of the dosage, subjects will remain on LZD treatment for 18 months after sputum culture conversion or until they can no longer tolerate therapy.
- Delayed Start Linezolid: Subjects will continue their existing regimen for 2 months after which LZD (600 mg once daily) will be added. After 2 consecutive AFB negative sputum smears (not to exceed 4 months of LZD therapy), subjects will be randomized to continue on 600 mg LZD once daily or to de-escalate to 300 mg once daily. Regardless of the dosage, subjects will remain on LZD treatment for 18 months after sputum culture conversion or until they can no longer tolerate therapy.
- Total: Total of all reporting groups
Arm/Group | Immediate Start Linezolid | Delayed Start Linezolid | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (11.2) | 40.4 (9.8) | 41.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Converted to Sputum Culture Negative in Each Arm, With Data Censored at 4 Months.
Time Frame: Sputum smear conversion or max 4 months after the start of Linezolid therapy.
Measure: Number; unit: participants
Arm/Group | Immediate Start Linezolid | Delayed Start Linezolid
Number analyzed (Participants) | 19 | 20
participants | 15 | 7

ADVERSE EVENTS:
Time Frame: Data were collected for the duration of the study subject's participation in the trial, up to 3 years. 39 subjects were included in the overall analysis but only 38 were at risk for AE because 1 subject did not receive LZD.
Description: AEs were collected on beginning treatment with LZD. AEs are not stratified by LZD dosage because all patients initiated LZD at 600 mg daily but then were subsequently randomized to either continue 600 mg or 300 mg daily. Thus a subject with AE on 300 mg likely reflects prior 600 mg dosing in addition to the current 300 mg dosing.
Groups:
- Clinically Significant AEs: All clinically significant adverse events, regardless of relationship to linezolid. This includes all SAEs, all AEs grade 3 and above, and all neuropathies grade 2 and above.
Arm/Group | Clinically Significant AEs
Serious Adverse Events (participants affected / at risk) | 25/38
Other Adverse Events (participants affected / at risk) | 24/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinically Significant AEs (N=38)
anemia (Blood and lymphatic system disorders) | 6 (7)
fever (Infections and infestations) | 1 (1)
esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hepatitis (Hepatobiliary disorders) | 3 (3)
hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (4)
neurologic reaction to psychotic drug (Nervous system disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 1 (1)
optic neuropathy (Eye disorders) | 7 (9)
peripheral neuropathy (Nervous system disorders) | 6 (6)
rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
vertigo (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinically Significant AEs (N=38)
cataract (Eye disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
hepatitis (Hepatobiliary disorders) | 1 (1)
hyperglycemia (Endocrine disorders) | 3 (3)
hyperuricemia (Musculoskeletal and connective tissue disorders) | 2 (2)
peripheral neuropathy (Nervous system disorders) | 15 (15)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes